CLINICAL TRIAL: NCT03453905
Title: Evaluation of the Ability of CT-based Finite Element Analysis (CTFEA) to Predict Fractures in Patients With Metastases: a Randomized Controlled Study.
Acronym: ZYCTFEA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0532-17-TLV
Record Dates: First submitted 2018-02-15; First posted 2018-03-05 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-02

CONDITIONS: Bone Neoplasm of Hip (Diagnosis); Orthopedic Disorder; Bone Metastases; Proximal Femoral Metaphyseal Abnormality
Keywords: CT-based Finite Element Analysis; Randomized Controlled Study; Preventive bone fixation; Randomized Controlled Trial
MeSH Terms: conditions — Disease; Musculoskeletal Diseases | interventions — Congresses as Topic

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to two arms and followed prospectively
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTFEA (Experimental): Decision on preventive surgery vs follow-up will be based on expert judgement, Mirels' score and CTFEA
  Interventions: Diagnostic Test: CTFEA
- Mirels (Other): Decision on preventive surgery vs follow-up will be based on expert judgement and Mirels' score
  Interventions: Other: Conventional decision algorithm

INTERVENTIONS:
Diagnostic Test: CTFEA — CT scans are used to generate a finite element model of patient-specific long bones. The bone model is loaded in stance position. Load based on patient's weight and the mechanical response, including the risk of fracture, is computed.
  Other Names: CT-based Finite Element Analysis
  Arms: CTFEA
Other: Conventional decision algorithm — Decision on surgery vs follow-up will be based on expert opinion and Mirels' score
  Other Names: Conventional
  Arms: Mirels

SUMMARY:
Patients with metastases to proximal femur, who are evaluated fr the risk of pathologic fracture in order to decide on preventive fixation vs follow-up constitute the study population. The patients will be randomized in two arms. First arm - the decision of treatment will rely on conventional decision algorithm including specialist judgement and Mirels' score. Second arm- the decision on treatment will be supported by CTFEA analysis of bone structure and quantitative simulation-based estimate of fracture risk, in addition to the conventional decision algorithm. Operation rates, pathologic fracture rates and additional secondary outcomes will be compared between the two study arms.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic bone disease of femur
2. Patients who undergo a CT scan (soft tissue kernel/filter, 120 kVp), and have at least 2/3 of both femurs visible in the CT scan. If CT scan is performed at the Sourasky medical center it must be according to the protocol in Appendix A.

Exclusion Criteria:

1. Ipsilateral previous surgery with or without implants
2. Low quality CT scan or CT does not include at least 2/3 of the femurs.
3. History of fractures, radiation or surgeries in lower limbs.
4. Inability to provide informed consent

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy hypothesis | four years
  To compare proportion of patients undergoing surgery in the treatment group vs the control group.

SECONDARY OUTCOMES:
Composite endpoint | 4 months
  pathological fracture during 4 months of follow up OR death within 30 days after prophylactic surgery in patients who underwent surgery OR surgical complications within 4 months of follow up: infection, re-operation, mechanical failure

OTHER OUTCOMES:
All-cause mortality | 4 years
  All-cause mortality
Number of patients who became unable to ambulate | 4 years
  Number of patients who became unable to ambulate for any reason. Inability to ambulate will be determined by an orthopedic surgeon from anamnesis and physical examination.
Number of participants who sustained a pathological fracture | 4 months
  Number of participants who sustained a pathological fracture. Diagnosis of pathological fracture will be determined by an orthopedic surgeon based on imaging.
Death | 30 days
  Death within 30 days after prophylactic surgery
Surgical complications | 4 months
  Infection, re-operation, mechanical failure within 4 months of follow up
Number of surgeries avoided | 4 months
  The number of surgeries "avoided" - presented only in the group of Intervention and only in patients without the safety endpoint within 4 months of follow up. Specifically, number of patients without the safety endpoint in whom a physician changed his/her decision to operate based on the CT-based FE analysis.
Agreement of two measures of fracture risk | One week
  Agreement between the pathological fracture risk estimated using Mirels' scale and the pathological fracture risk CT-based FE simulation analysis. Risk levels determined by either of the estimates: low, medium, high
Patients who denied surgery | 4 months
  Number of patients who did not undergo a prophylactic surgery, in whom the CT-based FE analysis showed a risk above moderate for fractures in future and who developed a fracture during the 4 months of follow-up - calculated in both study groups.
Complications that could be prevented by CTFEA | One month
  Number of patients who underwent a prophylactic surgery, in whom the CT-based FE analysis showed a mild-moderate risk of a fracture and who devel-oped a complication (as defined in a composite safety endpoint) - calculated in both study groups

CONTACTS AND LOCATIONS:
Overall Officials: Amir Sternheim, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center

IPD SHARING:
Plan to Share IPD: No
The individual participant data will remain in TLVMC and will not be shared

REFERENCES:
- [Background] Bickels J, Dadia S, Lidar Z. Surgical management of metastatic bone disease. J Bone Joint Surg Am. 2009 Jun;91(6):1503-16. doi: 10.2106/JBJS.H.00175. PMID 19487532
- [Background] Mirels H. Metastatic disease in long bones. A proposed scoring system for diagnosing impending pathologic fractures. Clin Orthop Relat Res. 1989 Dec;(249):256-64. PMID 2684463
- [Background] Goodheart JR, Cleary RJ, Damron TA, Mann KA. Simulating activities of daily living with finite element analysis improves fracture prediction for patients with metastatic femoral lesions. J Orthop Res. 2015 Aug;33(8):1226-34. doi: 10.1002/jor.22887. Epub 2015 May 21. PMID 25761000
- [Background] Yosibash Z, Trabelsi N, Milgrom C. Reliable simulations of the human proximal femur by high-order finite element analysis validated by experimental observations. J Biomech. 2007;40(16):3688-99. doi: 10.1016/j.jbiomech.2007.06.017. Epub 2007 Aug 13. PMID 17706228
- [Background] Trabelsi N, Yosibash Z, Wutte C, Augat P, Eberle S. Patient-specific finite element analysis of the human femur--a double-blinded biomechanical validation. J Biomech. 2011 Jun 3;44(9):1666-72. doi: 10.1016/j.jbiomech.2011.03.024. Epub 2011 Apr 15. PMID 21497354
- [Background] Yosibash Z, Plitman Mayo R, Dahan G, Trabelsi N, Amir G, Milgrom C. Predicting the stiffness and strength of human femurs with real metastatic tumors. Bone. 2014 Dec;69:180-90. doi: 10.1016/j.bone.2014.09.022. Epub 2014 Oct 2. PMID 25284156
- [Background] Benca E, Patsch JM, Mayr W, Pahr DH, Windhager R. The insufficiencies of risk analysis of impending pathological fractures in patients with femoral metastases: A literature review. Bone Rep. 2016 Mar 2;5:51-56. doi: 10.1016/j.bonr.2016.02.003. eCollection 2016 Dec. PMID 28326347
- [Background] Nazarian A, Entezari V, Zurakowski D, Calderon N, Hipp JA, Villa-Camacho JC, Lin PP, Cheung FH, Aboulafia AJ, Turcotte R, Anderson ME, Gebhardt MC, Cheng EY, Terek RM, Yaszemski M, Damron TA, Snyder BD. Treatment Planning and Fracture Prediction in Patients with Skeletal Metastasis with CT-Based Rigidity Analysis. Clin Cancer Res. 2015 Jun 1;21(11):2514-9. doi: 10.1158/1078-0432.CCR-14-2668. Epub 2015 Feb 27. PMID 25724521